CLINICAL TRIAL: NCT00854802
Title: A Multicentre, Randomised, Double-blind, Placebo-controlled, Parallel-group Phase II Study on the Efficacy and Safety of Debio 025 Combined With Peg-IFNα2a and Ribavirin in Treatment naïve Chronic Hepatitis C Genotype 1 Patients
Brief Title: A Study of Debio 025 (Alisporivir) Combined With Peg-IFNα2a and Ribavirin in Treatment naïve Chronic Hepatitis C Genotype 1 Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Debiopharm International SA (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Debio 025-HCV-205; 2008-004605-34 (EudraCT Number); CDEB025A2205 (Other: Sponsor Code)
Record Dates: First submitted 2009-03-02; First posted 2009-03-03 (Estimated); Last update posted 2016-02-17 (Estimated); Status verified 2016-02

CONDITIONS: Chronic Hepatitis C
Keywords: Hepatitis; Hepatitis C
MeSH Terms: conditions — Hepatitis C, Chronic; Hepatitis; Hepatitis C | interventions — alisporivir; peginterferon alfa-2a; Ribavirin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Debio 025 600 mg + peg-IFNα2a + ribavirin - 48 weeks (Experimental): Participants receive Debio 025 600 mg orally twice daily for 7 days (loading dose) followed by Debio 025 600 mg orally once daily for 47 weeks + peg-IFNα2a 180 µg subcutaneously (sc) once weekly for 48 weeks + ribavirin 1000 or 1200 mg (weight based) orally daily for 48 weeks.
  Interventions: Drug: Debio 025; Drug: Peg-IFNα2a; Drug: Ribavirin
- Debio 025 600 mg + peg-IFNα2a + ribavirin - 24 weeks (Experimental): Participants receive Debio 025 600 mg orally twice daily for 7 days (loading dose) followed by Debio 025 600 mg orally once daily for 23 weeks + peg-IFNα2a 180 µg sc once weekly for 24 weeks + ribavirin 1000 or 1200 mg (weight based) orally daily for 24 weeks.
  Interventions: Drug: Debio 025; Drug: Peg-IFNα2a; Drug: Ribavirin
- Debio 025 600 mg + peg-IFNα2a + ribavirin - 24 or 48 weeks (Experimental): Participants receive Debio 025 600 mg orally twice daily for 7 days (loading dose) followed by Debio 025 600 mg orally once daily for 23 or 47 weeks + peg-IFNα2a 180 µg sc once weekly for 24 or 48 weeks + ribavirin 1000 or 1200 mg (weight based) orally daily for 24 or 48 weeks. Participants who achieve a rapid viral response, defined as having undetectable hepatitis C virus RNA at week 4, are treated for 24 weeks; other patients are treated for 48 weeks.
  Interventions: Drug: Debio 025; Drug: Peg-IFNα2a; Drug: Ribavirin
- Debio 025 placebo + peg-IFNα2a + ribavirin - 48 weeks (Placebo Comparator): Participants receive Debio 025 placebo orally twice daily for 7 days followed by Debio 025 placebo orally once daily for 47 weeks + peg-IFNα2a 180 µg subcutaneously (sc) once weekly for 48 weeks + ribavirin 1000 or 1200 mg (weight based) orally daily for 48 weeks.
  Interventions: Drug: Peg-IFNα2a; Drug: Ribavirin; Drug: Debio 025 placebo

INTERVENTIONS:
Drug: Debio 025 — Debio 025 supplied in soft gel capsules
  Other Names: Alisporivir
  Arms: Debio 025 600 mg + peg-IFNα2a + ribavirin - 24 or 48 weeks; Debio 025 600 mg + peg-IFNα2a + ribavirin - 24 weeks; Debio 025 600 mg + peg-IFNα2a + ribavirin - 48 weeks
Drug: Peg-IFNα2a — Peg-IFNα2a supplied in pre-filled syringes
  Other Names: Pegasys
Drug: Ribavirin — Ribavirin supplied in tablets
  Other Names: Copegus; Rebetol; Ribasphere; Vilona; Virazole
Drug: Debio 025 placebo — Debio 025 placebo supplied in soft gel capsules
  Arms: Debio 025 placebo + peg-IFNα2a + ribavirin - 48 weeks

SUMMARY:
The purpose of this study is to compare several Debio 025 (alisporivir)/peg-IFNα2a/ribavirin triple therapies with the current standard of care (SOC) in treatment naïve chronic hepatitis C genotype 1 patients.

DETAILED DESCRIPTION:
This is an international, multicentre, randomised, double-blind, placebo-controlled, 4-arm, parallel-group, multiple dose phase II study comparing 3 Debio 025 (alisporivir)/peg-IFNα2a/ribavirin regimens to SOC treatment in treatment naïve chronic HCV genotype 1 patients.

Patients are randomised into 1 of 4 arms receiving either Debio 025/peg-IFNα2a/ribavirin triple therapy for a fixed treatment duration of 48 weeks (Treatment A) or 24 weeks (Treatment B), Debio 025/peg-IFNα2a/ribavirin triple therapy for a response-based treatment duration of 24 or 48 weeks (Treatment C), or blinded SOC treatment for 48 weeks (Treatment D). Follow-up is 24 weeks in all treatment arms.

ELIGIBILITY:
Inclusion Criteria:

* Males or females aged ≥ 18 and ≤ 65 years.
* Body mass index (BMI) ≥ 18 and ≤ 32 kg/m^2.
* Hepatitis B surface antigen (HbsAg) negative and HIV-1 negative.
* Serological diagnosis of chronic hepatitis C viral infection genotype 1 for > 6 months.
* Chronic liver disease consistent with chronic hepatitis C infection on a biopsy or FibroScan® obtained within the past 24 months (36 months for patients with incomplete/transition to cirrhosis).
* Previously untreated for hepatitis C virus (HCV) infection (approved or investigational drug).
* Plasma HCV RNA level lower limit ≥ 100 IU/ml assessed by quantitative polymerase chain reaction (qPCR) or equivalent; no upper limit.
* Neutrophil count ≥ 1500/µL; hemoglobin (Hb) ≥ 12g/dL for females and ≥ 13g/dL for males; platelets ≥ 90,000/µL.
* Patients with incomplete/transition to cirrhosis on biopsy or an elasticity score between 9.5 and 14 kPa on FibroScan must have an abdominal ultrasound (US), computed tomographic (CT) scan, or magnetic resonance imaging (MRI) scan without evidence of hepatocellular carcinoma (within 2 months prior to randomisation) and a serum alpha-foetoprotein (AFP) < 100 ng/mL.
* Aspartate aminotransferase (ASAT) and alanine aminotransferase (ALAT) < 5 times the upper limit of normal.
* Normal or compensated liver function and absence of complicated portal hypertension as documented by the following:

  * No history of bleeding oesophageal varices;
  * Absence of ascites;
  * Absence of encephalopathy;
  * Albumin ≥ 35 g/L;
  * Total bilirubin ≤ 1.8 mg/dL (≤ 30 µmol/L);
  * Prothrombin (INR ≤ 1.5).
* Creatinine clearance > 50 mL/min.
* Thyroid stimulating hormone (TSH) within normal range;
* All patients should be informed about Debio 025 and ribavirin foetotoxicity:

  * Females may participate if they are surgically sterile or post-menopausal. Pre-menopausal females may participate if they use 2 reliable contraceptive methods (oral contraceptive + barrier method). The contraceptive regimen must be maintained during the treatment period and for 4 months after the last Debio 025 or ribavirin dose.
  * Male patients must be surgically sterile or use 2 reliable contraceptive methods (oral contraceptive + barrier method). The contraceptive regimen must be maintained during the treatment period and for 7 months after the last Debio 025 or ribavirin dose.
* Signed informed consent before any study procedures.
* Negative pregnancy test within one week of first investigational product administration for female patients of child bearing potential.

Exclusion Criteria:

* Treatment with any investigational drug within 6 months prior to the first dose of investigational product.
* HCV genotype different from genotype 1.
* Any previous HCV treatment (approved or investigational).
* Histologic evidence of complete hepatic cirrhosis (including compensated cirrhosis) based on a previous liver biopsy (if available).
* Ongoing or recent use of any other medication (including over the counter medication and herbal products) within 2 weeks before study start or within 5 drug half-lives of that medication (whichever is longer) that are known inhibitors/inducers of cytochrome P450 (CYP450) 3A, substrates of P-glycoprotein 1 (P-gP), or substrates/inhibitors of organic anion-transporting polypeptides (OATP), multidrug resistance-associated protein 2 (MRP2), or bile salt export pump (BSEP) and are mentioned in the list of unauthorised medications;
* Any medical contraindications to peg-IFNα2a and/or ribavirin treatment;
* Any other cause of relevant liver disease other than HCV including but not limited to hepatitis B virus (HBV), drug- or alcohol-related cirrhosis, autoimmune hepatitis, haemochromatosis, Wilson's disease, nonalcoholic steatohepatitis (NASH), primary sclerosing cholangitis (PSC), or primary biliary cirrhosis (PBC).
* Any other condition which, in the opinion of the Investigator, would make the patient unsuitable for enrollment or could interfere with the patient participating in and completing the study. Patients with risk factors (hypertension or diabetes) need to have an ophthalmologic investigation (including fundoscopy).
* History of moderate, severe, or uncontrolled psychiatric disease, especially depression, including a history of hospitalisation or prior suicidal attempt.
* Uncontrolled arterial hypertension, ie, patients with systolic BP ≥ 160 mmHg and/or diastolic BP ≥ 100 mmHg.
* History of pancreatitis, uncontrolled diabetes mellitus, or retinopathy.
* Anti-nuclear antibody (ANA) titre > 1:640 at screening and/or evidence of autoimmune hepatitis on liver biopsy.
* Alcohol consumption > 20 g/day for females and > 30 g/day for males.
* History of major organ transplantation with an existing functional graft.
* Pregnancy or lactation.
* Haemoglobinopathies (thalassaemia major, sickle cell anaemia or drepanocytosis).
* Familial history of severe neonatal cholestasis or pregnancy cholestasis.
* Evidence of an active or suspected cancer, or a history of malignancy where the risk of recurrence is ≥ 20% within 2 years.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 290 (Actual)
Dates: Start 2009-01; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Percentage of participants achieving sustained viral response (SVR) 72 weeks after treatment start | 72 weeks after treatment start
  SVR is defined as hepatitis C virus (HCV) RNA < 10 IU/mL (undetectable).

SECONDARY OUTCOMES:
Percentage of participants achieving a rapid viral response (RVR) after 4 weeks of treatment | 4 weeks after treatment start
  RVR is defined as HCV RNA level < 10 IU/mL after 4 weeks of treatment.
Percentage of participants achieving a complete early viral response (cEVR) after 12 weeks of treatment | 12 weeks after treatment start
  cEVR is defined as HCV RNA level < 10 IU/mL after 12 weeks of treatment.
Percentage of participants achieving an early viral response (EVR) after 12 weeks of treatment | 12 weeks after treatment start
  EVR is defined as a decrease from baseline of the HCV RNA level by > 2 log10 or undetectable (< 10 UI/mL) after 12 weeks of treatment.
Percentage of participants achieving an end-of-treatment response (ETR) at treatment end | at end of treatment (Week 28 or Week 52)
  ETR is defined as HCV RNA level < 10 IU/mL at the end of treatment (Week 24 or Week 48).
Percentage of participants achieving a sustained viral response 12 weeks after the end of treatment (SVR 12) | 12 weeks after end of treatment (Week 40 or Week 64)
  SVR 12 is defined as HCV RNA level < 10 IU/mL 12 weeks after the end of treatment (Week 40 or Week 64).
Percentage of participants with sustained viral response 24 weeks after the end of treatment (SVR 24) | 24 weeks after end of treatment (Week 52 or Week 76
  SVR 24 is defined as HCV RNA level < 10 IU/mL 24 weeks after the end of treatment (Week 52 or Week 76).

CONTACTS AND LOCATIONS:
Overall Officials: Rafael Crabbé, MD, Study Director — Debiopharm International SA
Locations (40):
- Belgium (2):
  - Cliniques Universitaires Saint-Luc, Brussels
  - UZ Gent, Ghent
- France (7):
  - C.H.U - Hôpital Henri-Mondor, Créteil
  - C.H.U de Lyon Hôpital de l'Hôtel Dieu, Lyon
  - Hôpital de l'Archet 2, Nice
  - C.H.U Hôpital Cochin, Paris
  - C.H.U - Hôpital Saint Antoine, Paris - Saint Antoine
  - Hôpital du Haut-Levêque - C.H.U de Bordeaux, Pessac
  - C.H.U de Nancy-Hôpital Brabois, Vandœuvre-lès-Nancy
- Germany (9):
  - Charité - Universitatsmedizin Berlin, Berlin
  - Universitätsklinikum Düsseldorf, Düsseldorf
  - Center for HIV and Hepatogastroenterology, Düsseldorf
  - Universitätsklinikum Essen, Essen
  - J.W. Goethe University Hospital, Frankfurt am Main
  - Albert-Ludwigs-Universität Freiburg, Universitätsk, Freiburg im Breisgau
  - Medizinische Hochschule Hannover, Hanover
  - Medizinische Universitätsklinik, Heidelberg
  - Johannes Gutenberg-Universitaet Mainz, Mainz
- Italy (5):
  - Policlinico S.Orsola Malpighi, Bologna
  - Mangiagalli e Regina Elena di Milano, Milan
  - Seconda Università di Napoli- Secondo Policlinico, Napoli
  - "Policlinico ""Paolo Giaccone"" dell'Università di, Palermo
  - Az. Osp. Universitaria S. Giovanni Battista, Torino
- Poland (7):
  - Wojewódzki Szpital Specjalistyczny im. K. Dluskieg, Bialystok
  - Wojewódzki Szpital Obserwacyjno-Zakazny im. Tadeus, Bydgoszcz
  - Szpital Specjalistyczny w Chorzowie, Chorzów
  - Wojewódzki Szpital Zespolony w Kielcach, Kielce
  - Krakowski Szpital Specjalistyczny im. Jana Pawla I, Krakow
  - Wojewódzki Szpital Specjalstyczny im. Wl. Biegansk, Lódz
  - Samodzielny Publiczny Zaklad Opieki Zdrowotnej Woj, Warsaw
- Romania (5):
  - Spitalul Clinic Colentina, Bucharest
  - Institutul Clinic Fundeni, Bucharest
  - Centrul de Diagnostic si Tratament Dr. Victor Babe, Bucharest
  - "Spitalul Clinic de Urgenta ""Prof. dr. Octavian F, Cluj-Napoca
  - Institutul de Gastroenterologie si Hepatologie, Iași
- Spain (5):
  - Hospital Universitari Vall d'Hebrón, Barcelona
  - Hospital Universitari Germans Trias i Pujol, Barcelona
  - Hospital Universitario de La Princesa, Madrid
  - Hospital Universitario Puerta de Hierro, Madrid
  - Hospital Universitario Nuestra Señora de Valme, Seville

REFERENCES:
- [Background] Paeshuyse J, Kaul A, De Clercq E, Rosenwirth B, Dumont JM, Scalfaro P, Bartenschlager R, Neyts J. The non-immunosuppressive cyclosporin DEBIO-025 is a potent inhibitor of hepatitis C virus replication in vitro. Hepatology. 2006 Apr;43(4):761-70. doi: 10.1002/hep.21102. PMID 16557546
- [Background] Inoue K, Umehara T, Ruegg UT, Yasui F, Watanabe T, Yasuda H, Dumont JM, Scalfaro P, Yoshiba M, Kohara M. Evaluation of a cyclophilin inhibitor in hepatitis C virus-infected chimeric mice in vivo. Hepatology. 2007 Apr;45(4):921-8. doi: 10.1002/hep.21587. PMID 17393519
- [Background] Flisiak R, Horban A, Gallay P, Bobardt M, Selvarajah S, Wiercinska-Drapalo A, Siwak E, Cielniak I, Higersberger J, Kierkus J, Aeschlimann C, Grosgurin P, Nicolas-Metral V, Dumont JM, Porchet H, Crabbe R, Scalfaro P. The cyclophilin inhibitor Debio-025 shows potent anti-hepatitis C effect in patients coinfected with hepatitis C and human immunodeficiency virus. Hepatology. 2008 Mar;47(3):817-26. doi: 10.1002/hep.22131. PMID 18302285
- [Background] Reesink HW, Zeuzem S, Weegink CJ, Forestier N, van Vliet A, van de Wetering de Rooij J, McNair L, Purdy S, Kauffman R, Alam J, Jansen PL. Rapid decline of viral RNA in hepatitis C patients treated with VX-950: a phase Ib, placebo-controlled, randomized study. Gastroenterology. 2006 Oct;131(4):997-1002. doi: 10.1053/j.gastro.2006.07.013. PMID 17030169
- [Background] Pawlotsky JM. Treatment of hepatitis C: don't put all your eggs in one basket! Gastroenterology. 2007 Apr;132(4):1611-5. doi: 10.1053/j.gastro.2007.03.014. No abstract available. PMID 17418174
- [Background] Dienstag JL, McHutchison JG. American Gastroenterological Association technical review on the management of hepatitis C. Gastroenterology. 2006 Jan;130(1):231-64; quiz 214-7. doi: 10.1053/j.gastro.2005.11.010. No abstract available. PMID 16401486
- [Background] Zeuzem S, Buti M, Ferenci P, Sperl J, Horsmans Y, Cianciara J, Ibranyi E, Weiland O, Noviello S, Brass C, Albrecht J. Efficacy of 24 weeks treatment with peginterferon alfa-2b plus ribavirin in patients with chronic hepatitis C infected with genotype 1 and low pretreatment viremia. J Hepatol. 2006 Jan;44(1):97-103. doi: 10.1016/j.jhep.2005.10.003. Epub 2005 Nov 7. PMID 16290907
- [Background] Watashi K, Hijikata M, Hosaka M, Yamaji M, Shimotohno K. Cyclosporin A suppresses replication of hepatitis C virus genome in cultured hepatocytes. Hepatology. 2003 Nov;38(5):1282-8. doi: 10.1053/jhep.2003.50449. PMID 14578868
- [Background] Watashi K, Ishii N, Hijikata M, Inoue D, Murata T, Miyanari Y, Shimotohno K. Cyclophilin B is a functional regulator of hepatitis C virus RNA polymerase. Mol Cell. 2005 Jul 1;19(1):111-22. doi: 10.1016/j.molcel.2005.05.014. PMID 15989969
- [Background] Rice CM, You S. Treating hepatitis C: can you teach old dogs new tricks? Hepatology. 2005 Dec;42(6):1455-8. doi: 10.1002/hep.20975. PMID 16317665
- [Background] Ishii N, Watashi K, Hishiki T, Goto K, Inoue D, Hijikata M, Wakita T, Kato N, Shimotohno K. Diverse effects of cyclosporine on hepatitis C virus strain replication. J Virol. 2006 May;80(9):4510-20. doi: 10.1128/JVI.80.9.4510-4520.2006. PMID 16611911
- [Background] Yang F, Robotham JM, Nelson HB, Irsigler A, Kenworthy R, Tang H. Cyclophilin A is an essential cofactor for hepatitis C virus infection and the principal mediator of cyclosporine resistance in vitro. J Virol. 2008 Jun;82(11):5269-78. doi: 10.1128/JVI.02614-07. Epub 2008 Apr 2. PMID 18385230
- See also: Study sponsor — http://www.debiopharm.com